CLINICAL TRIAL: NCT01639651
Title: Principal Investigator
Brief Title: The Acute Effect of a Mobilization With Movement Technique to Improve Internal Rotation of the Shoulder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Renato Rozenblit Soliaman, The Acute Effect of a Mobilization With Movement Technique to Improve Internal Rotation of the Shoulder: a Randomized Controlled Trial, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02195112.7.0000.5505
Record Dates: First submitted 2012-07-09; First posted 2012-07-13 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Disorder of Shoulder; Other Musculoskeletal Disorder; Contracture
Keywords: Physical Therapy; Glenohumeral Internal Rotation Deficits; Joint Mobilization; Posterior capsule; Capsular contracture
MeSH Terms: conditions — Contracture | interventions — Control Groups; Movement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Posterior capsule stretching
- Mobilization Group (Experimental)
  Interventions: Other: Mobilization with movement

INTERVENTIONS:
Other: Posterior capsule stretching — Control group that will be submitted for an evaluation of shoulder range of motion (internal/external rotation)for both limbs, upper limb active movements to warm-up (five minutes), posterior capsule stretching (Cross-body stretch for 3 sets of 30 seconds) and revaluation immediately post-intervention and four weeks post-intervention.
  Other Names: Control group
  Arms: Control Group
Other: Mobilization with movement — Mobilization group that will be submitted for an evaluation of shoulder range of motion (internal/external rotation) for both limbs, upper limb active movements to warm-up (five minutes), posterior capsule stretching (Cross-body stretch for 3 sets of 30 seconds) plus a mobilization with movement to improve internal rotation of the dominant shoulder (three sets of 10 repetitions)and revaluation immediately post-intervention and four weeks post-intervention.
  Other Names: Experimental Group
  Arms: Mobilization Group

SUMMARY:
For many years researchers have been documented that the shoulder of the throwing athlete acquires a increase in external rotation of the dominant limb compared to the contralateral side.This fact is followed with a loss of the internal rotation of the shoulder, which is related with a higher rate of injuries in this joint and it´s known as Glenohumeral Internal Rotation Deficit (GIRD).

Among the approaches for this condition the literature is inconclusive due to the low methodological quality of clinical trials made,however, the manual therapy has been used with success to relief the pain and restore the range of motion.

The purpose of this study is to analyse the effectiveness of a mobilization with movement technique to improve the internal rotation of the shoulder in throwing athletes with GIRD.

It will be a randomized controlled trial with the CONSORT bases with 40 participants that will be divided into two groups:

* Control group that will be submitted for an evaluation of shoulder range of motion (internal/external rotation)of both limbs, upper limb active movements to warm-up (five minutes), posterior capsule stretching (Cross-body stretch for 3 sets of 30 seconds) and revaluation immediately post-intervention and four weeks post-intervention.
* Mobilization group that will be submitted for an evaluation of shoulder range of motion (internal/external rotation)of both limbs, upper limb active movements to warm-up(five minutes), posterior capsule stretching (Cross-body stretch for 3 sets of 30 seconds) plus a mobilization with movement technique to improve internal rotation of the dominant shoulder (three sets of 10 repetitions)and revaluation immediately post-intervention and four weeks post-intervention.

To evaluate the range of movement it will be use a standard goniometer with an attached customizes bubble inclinometer to ensure proper perpendicular alignment of the goniometer to the ground.

The investigators hypothesis is that both group will have improvements in the internal rotation of the dominant shoulder, however, the mobilization group will have a statistically significant difference compared to control group immediately post-intervention. Four weeks post-intervention this difference will equalize, because of the only intervention applied.

Results will be expressed as hazard ratios (HR) with their respective confidence intervals at 95% and adopting α = 0.05. All analyzes will be performed by SPSS version 17.0

ELIGIBILITY:
Inclusion Criteria:

* Athletes that practice at least 10 hours of throwing sports.
* Glenohumeral internal rotation deficits of the dominant shoulder compare to the non-dominant limb.
* Agree to participate and signing the informed consent approved for the Federal University of São Paulo ethics committee.

Exclusion Criteria:

* Previous surgeries of the shoulders.
* Unable to perform the evaluation or treatment due to pain.
* Performing physical therapy treatment.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Analyse the effectiveness of a mobilization with movement technique to improve internal rotation of the shoulder in throwers athletes with GIRD | Immediately post-intervention and four weeks post-intervention
  The 40 patients will be divided in two groups of 20. Both will perform a evaluation of the internal and external rotation of the shoulders to determine the individual internal rotation deficit of the dominant shoulder compared to the contralateral side. One group (Control) will perform what the literature recommends (Stretch of the posterior capsule), and the other group (Mobilization) will add to the control intervention a mobilization with movement technique to improve the internal rotation deficit which was identified previously.

CONTACTS AND LOCATIONS:
Overall Officials: Renato R Soliaman, Principal Investigator — Centro de Traumatologia do Esporte - CETE
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil